CLINICAL TRIAL: NCT05213156
Title: Concentration of Ofloxacin Into the Aqueous Humour of Patients After Topical Instillation According to the Severity of Dry Eye Disease
Brief Title: Concentration of Ofloxacin Into the Aqueous Humour of Patients With Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Collaborators: University of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Screening
Other Study IDs: 1094/31-12-18
Record Dates: First submitted 2021-12-23; First posted 2022-01-28 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Disease
Keywords: Inflammation; Dry Eye Disease; Therapeutics; Topical Application; Aqueous Humour
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants were didvided in three groups: the control group, those who suffer from severe Dry Eye Disease and all other patients with Dry Eye Disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients without Dry Eye Disease (Active Comparator): Control Group
  Interventions: Drug: Oxatrex
- Patients with Dry Eye Disease, except the severe Dry Eye Disease (Experimental): non severe Dry Eye Disease
  Interventions: Drug: Oxatrex
- Patients with severe Dry Eye Disease (Experimental): severe Dry Eye Disease
  Interventions: Drug: Oxatrex

INTERVENTIONS:
Drug: Oxatrex — 0.3% ofloxacin eye drops in single doses

SUMMARY:
After topical installation of one drop of 0.3% commercially available ofloxacin (Oxatrex®) four times at intervals of 15min in catarract patients with Dry Eye Disease, aqueous humour samples will be collected intraoperatively, one hour after the last installation. Concentration of ofloxacin in aqueous humour will be measured by HPLC-MS/MS.

DETAILED DESCRIPTION:
Patients will be categorized into three Groups, according to DED severity. Group I comprises of subjects without DED, Group II of patients are evaluated as non-severe DED, and Group III consists of patients suffering from severe DED.

The day before cataract surgery will be performed patient examination, during standard cataract preoperative evaluation. Briefly, symptom-based assessment will be delivered by scoring the Ocular Surface Disease Index (OSDI) questionnaire, and evaluation of ocular surface damage will be performed by corneal fluorescein staining using the Oxford scale.

Before surgery, patients will be assigned to receive one drop of commercially available topical ofloxacin solution 0.3% at monodoses without preservatives (Oxatrex, Zwitter Pharmaceuticals, Greece) four times at fifteen minutes intervals starting 2 hours before surgery. The eye drops will be applied in the middle of the inferior lower fornix. Patients who miss any of the 4 doses will be excluded from the study. Aqueous humor will be collected after 1 hour of the last administration, intraoperatively, at the beginning of cataract surgery.

A paracentesis track will be made with a 15ᵒ superblade, a 30G cannula, connected to a tuberculin syringe, will be inserted into the A/C and approximately 50 μL of aqueous humor will be withdrawn. AqH samples will be collected in an Eppendorf tube. All samples will kept frozen at -20ᵒC.

Ofloxacin concentrations will be determined by HPLC-MS/MS.

DED severity, symptoms (Ocular Surface Disease Index) and signs (corneal staining using the Oxford score) will be correlated to ofloxacin's concentration in the AqH.

ELIGIBILITY:
Inclusion Criteria:

* cataract surgery
* willing to participate

Exclusion criteria:

* presence of exfoliation material within the anterior segment of the eye
* pigment dispersion syndrome
* anterior chamber angle < 20ᵒ
* other ocular pathology than cataract
* abnormal eyelid function
* diabetes mellitus, renal or hepatic failure
* chronic topical ocular treatment
* systematic antibiotic treatment
* allergy to fluoroquinolone antibiotics
* contact lens use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
DED severity | One day prior to cataract surgery, from 09:00am to 12:00pm
  DED severity will be determined during preoperative cataract evaluation.
Concentration of ofloxacin in the aqueous humour | Beginning of the cataract surgery, from 08:30am to 12:30pm
  After topical instillation of ofloxacin eye drops, aqueous humor samples will be collected intraoperatively and ofloxacin concentration will be determined by HPLC-MS/MS.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | One day prior to cataract surgery, from 09:00am to 12:00pm
  Scoring of the OSDI questionnaire.
Corneal staining | One day prior to cataract surgery, from 09:00am to 12:00pm
  Εvaluation of ocular surface damage by corneal fluorescein staining using the Oxford scale.

CONTACTS AND LOCATIONS:
Overall Officials: Constantine D. Georgakopoulos, MD, PhD, Study Director — University Hospital of Patras
Locations (1):
- Department of Ophthalmology, General University Hospital of Patras, Pátrai, Achaea, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baudouin C, Aragona P, Van Setten G, Rolando M, Irkec M, Benitez del Castillo J, Geerling G, Labetoulle M, Bonini S; ODISSEY European Consensus Group members. Diagnosing the severity of dry eye: a clear and practical algorithm. Br J Ophthalmol. 2014 Sep;98(9):1168-76. doi: 10.1136/bjophthalmol-2013-304619. Epub 2014 Mar 13. PMID 24627252
- [Background] Perez VL, Stern ME, Pflugfelder SC. Inflammatory basis for dry eye disease flares. Exp Eye Res. 2020 Dec;201:108294. doi: 10.1016/j.exer.2020.108294. Epub 2020 Oct 8. PMID 33039458
- [Background] Agrahari V, Mandal A, Agrahari V, Trinh HM, Joseph M, Ray A, Hadji H, Mitra R, Pal D, Mitra AK. A comprehensive insight on ocular pharmacokinetics. Drug Deliv Transl Res. 2016 Dec;6(6):735-754. doi: 10.1007/s13346-016-0339-2. PMID 27798766
- [Background] Barar J, Javadzadeh AR, Omidi Y. Ocular novel drug delivery: impacts of membranes and barriers. Expert Opin Drug Deliv. 2008 May;5(5):567-81. doi: 10.1517/17425247.5.5.567. PMID 18491982
- [Background] Gatti G, Panozzo G. Effect of inflammation on intraocular penetration of intravenous ofloxacin in albino rabbits. Antimicrob Agents Chemother. 1995 Feb;39(2):549-52. doi: 10.1128/AAC.39.2.549. PMID 7726531
- [Background] Ozturk F, Kortunay S, Kurt E, Inan UU, Ilker SS, Basci N, Bozkurt A. The effect of long-term use and inflammation on the ocular penetration of topical ofloxacin. Curr Eye Res. 1999 Dec;19(6):461-4. doi: 10.1076/ceyr.19.6.461.5277. PMID 10550786
- [Background] Ozturk F, Kurt E, Inan UU, Kortunay MC, Ilker SS, Basci NE, Bozkurt A. Penetration of topical and oral ofloxacin into the aqueous and vitreous humor of inflamed rabbit eyes. Int J Pharm. 2000 Aug 25;204(1-2):91-5. doi: 10.1016/s0378-5173(00)00482-8. PMID 11011990